CLINICAL TRIAL: NCT03893916
Title: MEG Versus EEG HR for the Localization of the Epileptogenic Zone as Part of the Pre-surgical Assessment of Epilepsy
Acronym: EPIMEEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0134; 2018-A02452-53 (Other: ANSM)
Record Dates: First submitted 2019-03-21; First posted 2019-03-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Drug-resistant Epilepsy; Candidates for Surgical Treatment; Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort (Experimental): MEG - EEG HR
  Interventions: Procedure: MEG - EEG HR

INTERVENTIONS:
Procedure: MEG - EEG HR — MEG : Magnetoencephalography is the study of the magnetic fields produced by the electrical activity of the brain.
  MEG signals are obtained while the patient is placed in a device specific to this technique. The latter comprises a recording chamber, recording sensors which are placed in a cryostat and an electronic measuring system. The magnetic fields are measured while the subject is placed in a shielded magnetic chamber protecting it from variations in the ambient magnetic field (displacement of metal masses, sector ...).
  EEG HR: High Resolution EEG is defined as the recording of cerebral electrical activity with 128 electroencephalographic electrodes and with high temporal resolution usually followed by the use of source localization tools. The HR EEG is therefore derived from standard EEG techniques, but requires a higher number of electrodes and the use of source localization tools.

SUMMARY:
Drug-resistant partial epilepsies are disabling diseases for which surgical treatment may be indicated. The determination of the area to be operated (or 'epileptogenic zone') is based on a bundle of clinical arguments and neuroimaging, having a direct impact on surgical success.

Epileptic patients have electrical abnormalities that can be detected with surface electrophysiological examinations such as surface EEG or MagnetoEncephalography (MEG). The intracerebral source of these abnormalities can be localized in the brain using source modeling techniques from MEG signals or EEG signals if a sufficient number of electrodes is used (> 100, so-called high EEG technique Resolution = EEG HR). EEG HR and MEG are two infrequent state-of-the-art techniques.

The independent contribution of EEG HR and MEG for the localization of the epileptogenic zone has been shown in several studies. However, several modeling studies have shown that MEG and EEG HR have a different detection capacity and spatial resolution depending on the cortical generators studied. Modeling studies suggest that MEG has better localization accuracy than EEG for most cortical sources.

No direct comparison of the locating value of MEG and EEG HR for the localization of the epileptogenic zone has been performed to date in a large-scale clinical study.

In this prospective study, 100 patients with partial epilepsy who are candidates for epilepsy surgery, and for some of them with intracranial EEG recording, will benefit from two advanced electrophysiological examinations including magnetoencephalographic recording (MEG). ) interictal electrophysiological abnormalities and high-resolution EEG recording (128 electrodes) in addition to the usual examinations performed as part of the pre-surgical assessment, prior to cortectomy and / or intracranial EEG recording.

Based on recent work conducted in humans, we postulate:

* that the MEG and the EEG HR make it possible to precisely determine the epileptogenic zone, by using two approaches of definition of the epileptogenic zone (zone operated in the cured patients, zone at the origin of the crises during the intracranial recordings), but that the MEG is a little more precise than the EEG HR for the determination of the epileptogenic zone (we will try to highlight a difference of about 10%)
* that the quantitative study of the complementarity between EEG HR and MEG for modeling sources of epileptic spikes will show an added value in the use of both methods compared to the use of only one of the two methods
* that it is possible to determine the epileptogenic zone by determining the MEG model zone having the highest centrality value (hub) within the intercritical network by studying networks using graph theory.

ELIGIBILITY:
Inclusion Criteria:

* patients with partial epilepsy for at least 2 years and for whom are decided and planned: either i) a surgical procedure to resect the epileptogenic zone without prior intracranial EEG recording either ii) an intracranial EEG record needed before a possible cortectomy procedure
* Routine scalp EEG revealing known paroxysmal interictal abnormalities (at least 5 points on a 20-minute plot performed less than 2 years before inclusion in the study)
* Patient giving written consent

Exclusion Criteria:

* patient aged over 60 or under 18
* patients with contraindications to brain MRI and MEG
* women of childbearing age for whom a urine pregnancy test performed during the first visit would detect a pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2029-04-25 (Estimated); Study Completion 2029-04-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for whom there will be a spatial congruence between the operated area and the area modeled in EEG HR and MEG, among the population of patients operated and cured | Month 12 after Surgery
  We will consider that it is congruent when the most likely source model will be located in the resected focus determined by the postoperative MRI. The clinical outcome of the patients will be assessed 1 year after the intervention according to the Engel classification. Patients with an Engel Grade 1 score will be considered cured.

SECONDARY OUTCOMES:
To compare the ability of EEG HR and MEG to localize the epileptogenic zone by considering the epileptogenic zone as the brain area involved in the beginning of the crisis in patients requiring intracranial EEG recording | Month 12 after Surgery
  Proportion of patients for whom there will be a spatial congruence between the epileptogenic zone defined by intracranial EEG recording and the modeled zone in EEG HR and MEG, among the population of operated and cured patients. The clinical outcome of the patients will be assessed 1 year after the intervention according to the Engel classification. Patients with an Engel Grade 1 score will be considered cured.
To evaluate the spatial congruence between the zones modeled by the MEG and the EEG HR and the resected brain zone in the group of the patients not cured | Month 12 after Surgery
  Proportion of patients for whom there will be a spatial congruence between the operated area and the modeled area in EEG HR and MEG in the group of operated and unhealed patients.
Study the complementarity of EEG HR and MEG for the localization of the epileptogenic zone | Month 12 after Surgery
  proportion of patients for whom there will be a spatial congruence between the operated area and the modeled area GET HR with a priori MEG and without bias MEG and the proportion of patients for whom there will be a spatial congruence between the operated area and the zone modeled in MEG with a priori EEG HR and without a priori EEG HR, among the population of patients operated and cured.
To study the localization value of MEG intercritical network analysis for the detection of the epileptogenic zone via graph theory | Month 12 after Surgery
  Proportion of patients for whom there will be a spatial congruence between the operated area and the MEG model zone having the highest centrality value (hub) within the interictal network, among the population of patients operated and cured

CONTACTS AND LOCATIONS:
Overall Officials: Julien JUNG, Dr, Study Chair — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No